CLINICAL TRIAL: NCT03036995
Title: Repigmentation Using Apremilast and Phototherapy In Diffuse VITILIGO RAPID VITILIGO
Brief Title: Repigmentation Using Apremilast and Phototherapy In Diffuse VITILIGO
Acronym: Rapid Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-PP-06
Record Dates: First submitted 2017-01-06; First posted 2017-01-31 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apremilast - Group A (Experimental): Patient will receive narrow UVB treatment and apremilast (2 tablets for day) during 24 weeks. If the patient is responder (response is defined as an increase of at least 30 % in the VASI score at W24 compare to Baseline), he will receive narrow UVB treatment according the and apremilast during 24 weeks.
  Interventions: Drug: Apremilast
- Placebo - Group B (Placebo Comparator): Patient will receive UVB treatment and placebo (2 tablets for day) during 24 weeks. If the patient is responder (response is defined as an increase of at least 30 % in the VASI score at W24 compare to Baseline), he will receive narrow UVB treatment and placebo during 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apremilast — Patient will receive narrow UVB treatment and apremilast (2 tablets for day) during 24 weeks. If the patient is responder (response is defined as an increase of at least 30 % in the VASI score at W24 compare to Baseline), he will receive narrow UVB treatment according the and apremilast during 24 weeks.
  Arms: Apremilast - Group A
Other: Placebo — Patient will receive narrow UVB treatment and placebo (2 tablets for day) during 24 weeks. If the patient is responder (response is defined as an increase of at least 30 % in the VASI score at W24 compare to Baseline), he will receive narrow UVB treatment according the and placebo during 24 weeks.
  Arms: Placebo - Group B

SUMMARY:
Vitiligo is a depigmentation disorder affecting 0.5 to 2% of the general population. It is an acquired pigmentary disorder of the skin and mucous membranes that is characterized by circumscribed, depigmented macules and patches. Apremilast is a phosphosdiesterase 4 (PDE4) inhibitor that showed efficacy and very good tolerance in rheumatoid arthritis and psoriasis. Apremilast induces a potent activation of the cyclic AMP (cAMP) pathway leading to anti-inflammatory effect by decreasing the response of Th1 and Th17 lymphocytes. Interestingly, the cAMP pathway is also well demonstrated to be the main pathway for promoting melanogenesis and for inducing the differentiation and the proliferation of melanocytes. The principal aims is to compare, after 24 weeks of treatment, the efficacy of Apremilast at the label dosage in combination therapy with narrow band UVB versus placebo therapy with narrow band UVB for repigmentation in patients with non-segmental vitiligo. Patients with non-segmental vitiligo with BSA > 10% and patient with Vitiligo stable or slowly progressive for 3 months , seeking for treatment in the Department of Dermatology, University Hospital of Nice, France will be recruited into the study. The Patients are seen in consultation by the investigator, selection criteria are checked. All patients will receive full body narrow UVB treatment, twice weekly sessions of narrow UVB for 24 weeks.

From W24 to W48

* All responders* will receive narrow UVB treatment according the French clinical use i.e.twice weekly sessions of narrowband UVB for 24 weeks.
* All responders* will be randomized to receive either apremilast** 30mg BID or placebo.

  * Response is defined as an increase of at least 30 % in the VASI score at W24 compare to baseline **Responders initially randomized in the placebo arm will benefit of the titration At week 24, the non responders patients will stop the treatment and the study after the 4 weeks observationnal follow-up (W28).

Observational Follow-up Phase - W48 to W52 Four-week Observational Follow-up Phase for all subjects who complete the study (responders and non responders) or discontinue the study early.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-segmental vitiligo affecting at least 10% of BSA since at least 3 months.
* Patient requiring a treatment by UVB
* For both female of childbearing potential and male patients: Use of an effective contraceptive method during the study period (see Annex 5 for details)
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted
* Able to adhere to the study visit schedule and other protocol requirements
* Patient registered to the French Social Security

Exclusion Criteria:

1. Segmental or mixed vitiligo
2. Other than vitiligo, history of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease.
3. Any condition which would place the subject at unacceptable risk if he/she were to participate in the study.
4. Any condition that confounds the ability to interpret data from the study.
5. Pregnant or breast feeding, pregnancy urinary tests will be performed (see Annex 5 for details about pregnancy testing and contraception)
6. History of allergy to any component of apremilast
7. History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease)
8. Active substance abuse or a history of substance abuse within 6 months prior to Screening
9. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed at least 4 weeks prior to Screening.
10. Malignancy or history of malignancy (except for treated [ie, cured] basal cell or squamous cell in situ skin carcinomas and treated [ie, cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence)
11. Evidence of skin conditions that would interfere with clinical assessments
12. Topical therapy within 2 weeks of randomization
13. Prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources
14. Prior treatment with apremilast
15. Use of phototherapy within 4 weeks prior to randomization (ie, UVB, PUVA)
16. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives,
17. Patients assessed to be uncooperative
18. Participants in other clinical studies
19. Vulnerable people: pregnant or breast-feeding women (an urinary pregnancy test will be realized in every visit), minors, adults under guardianship or guardianship, deprived of freedom
20. Patient with a rare hereditary disease such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption syndrome
21. Patient with severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Score VASI | at 24 weeks
  Efficacy will be evaluated using the Vitiligo Area Scoring Index (VASI)

SECONDARY OUTCOMES:
Score VETF | at 24 weeks
  Efficacity will be also evaluated using the Vitiligo European Task Score (VETF)
Score VE | at 24 weeks
  Efficacy will be also evaluated using the Vitiligo Extent Score (VES)

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice - Dermatologie - Hôpital Archet, Nice, Alpes-Maritimes, France

REFERENCES:
- [Derived] Khemis A, Fontas E, Moulin S, Montaudie H, Lacour JP, Passeron T. Apremilast in Combination with Narrowband UVB in the Treatment of Vitiligo: A 52-Week Monocentric Prospective Randomized Placebo-Controlled Study. J Invest Dermatol. 2020 Aug;140(8):1533-1537.e2. doi: 10.1016/j.jid.2019.11.031. Epub 2020 Jan 29. PMID 32004567